CLINICAL TRIAL: NCT00892138
Title: Mindfulness Training for Stress Management: A Two-centre Randomised Controlled Study of Medical and Psychology Students With Long-term Follow up
Brief Title: Mindfulness Training for Stress Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Norwegian Knowledge Centre for the Health Services (Other Government)
Collaborators: University of Oslo (Other); University of Tromso (Other); Norwegian Medical Association (Other)
Responsible Party: Principal Investigator, Michael de Vibe, Senior Advisor, Norwegian Knowledge Centre for the Health Services
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 08/4352 Norw Medical Assoc
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Psychological Distress
Keywords: mindfulness training; medical students; psychology students; stress management; personal development; stress
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness training (Experimental): Mindfulness training
  Interventions: Behavioral: Mindfulness training
- Control (No Intervention): Study program as usual

INTERVENTIONS:
Behavioral: Mindfulness training — 7 week course modeled on MBSR according to Kabat-Zinn
  Other Names: Mindfulness-Based Stress Reduction
  Arms: Mindfulness training

SUMMARY:
This study will assess the short and long term effects of a group-based mindfulness programme (Mindfulness-Based Stress Reduction, MBSR) on first year medical and psychology students at the Universities of Oslo and Tromso.

The primary outcome variables are mental distress, student stress and subsequent work stress, subjective wellbeing, empathy, mindfulness and spirituality. The investigators will also study explanatory moderator and mediator variables.

The study will be a two-centre randomized controlled study involving 288 medical and psychology students from the University of Oslo and from the University of Tromso. The sample size calculation is based on a reduction in mental distress and perceived medical/psychology school stress of 20% in the intervention group. The control group will not receive an intervention. After the initial seven week course (taking place in 2009 and 2010) the intervention group will receive a follow-up session of 1.5 hours twice a year throughout their study course of 5-6 years. The follow-up period will last until 1 year after graduation in the Oslo cohort and until 3 years after graduation in the Tromso cohort.

ELIGIBILITY:
Inclusion Criteria:

* All students in term 3 of their medical and psychology study at the University of Oslo in the autumn of 2009, and spring of 2010.
* All students in term 3 of their medical and psychology study at the University of Tromso in the autumn of 2010, and autumn of 2011.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2009-09; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
The primary outcome variables are mental distress (GHQ12, SCL5 and MBI), student stress (PMSS) and subsequent work stress, subjective wellbeing (SWB), empathy (JPSE), mindfulness (FFMS) | 9 years
  The following predictor variables will be measured: Coping (WCCL), Regulatory focus, Personality (BCI), Perceived social support, Life events

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - University of Oslo, Oslo
  - University of Tromso, Tromsø

REFERENCES:
- [Derived] Kunzler AM, Helmreich I, Konig J, Chmitorz A, Wessa M, Binder H, Lieb K. Psychological interventions to foster resilience in healthcare students. Cochrane Database Syst Rev. 2020 Jul 20;7(7):CD013684. doi: 10.1002/14651858.CD013684. PMID 32691879
- [Derived] de Vibe M, Solhaug I, Rosenvinge JH, Tyssen R, Hanley A, Garland E. Six-year positive effects of a mindfulness-based intervention on mindfulness, coping and well-being in medical and psychology students; Results from a randomized controlled trial. PLoS One. 2018 Apr 24;13(4):e0196053. doi: 10.1371/journal.pone.0196053. eCollection 2018. PMID 29689081
- [Derived] de Vibe M, Solhaug I, Tyssen R, Friborg O, Rosenvinge JH, Sorlie T, Bjorndal A. Mindfulness training for stress management: a randomised controlled study of medical and psychology students. BMC Med Educ. 2013 Aug 13;13:107. doi: 10.1186/1472-6920-13-107. PMID 23941053